CLINICAL TRIAL: NCT04060316
Title: Efficacy, Safety, and Tolerability of Adjuvant GLS-1200 Topical Nasal Spray in the Prevention of Acute Rhinosinusitis Following Functional Endoscopic Sinus Surgery (FESS)
Brief Title: GLS-1200 Topical Nasal Spray to Prevent Sinusitis After Endoscopic Sinus Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: GeneOne Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: T2R-001
Record Dates: First submitted 2019-08-13; First posted 2019-08-19 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Sinusitis Chronic
Keywords: Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GLS-1200 (Experimental): 3 ml of GLS-1200 (1 mg/ml in 0.9% saline)
  Interventions: Drug: GLS-1200
- Sterile Saline (Placebo Comparator): 3 ml of 0.9% saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLS-1200 — GLS-1200 is given as a nasal spray using an atomizer
  Arms: GLS-1200
Drug: Placebo — Placebo is given as a nasal spray using an atomizer
  Other Names: Sterile Saline
  Arms: Sterile Saline

SUMMARY:
This clinical trial will evaluate the safety, tolerability and effectiveness of GLS-1200 nasal spray in addition to the standard of care after endoscopic sinus surgery in people with chronic sinusitis.

DETAILED DESCRIPTION:
Subjects will be assigned to treatment via nasal spray with either GLS-1200 or placebo in blinded manner in a 2:1 ratio. Treatment will commence 1 week post-operatively and continue for 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older;
* Able to provide informed consent
* Able and willing to comply with study procedures
* Elective FESS
* Able and willing to utilize an approved form of pregnancy prevention for women of child bearing potential

Exclusion Criteria:

* Pregnancy or documentation of pregnancy by pre-operative pregnancy test
* History of primary ciliary dyskinesia
* Known allergy to quinine, quinidine or mefloquine
* Know latex allergy
* History of hematologic malignancy
* History of bone marrow transplantation
* Current or planned chemotherapy treatment for hematologic or solid tumor during study period
* FESS performed non-electively and /or in preparation for decontamination of the sinuses related to cystic fibrosis or in preparation for chemotherapy, solid organ transplantation, or bone marrow transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Safety measures: treatment emergent adverse events by group will be summarized as frequencies by severity and relationship to treatment | Post-op through week 16 post-FESS
Assess the incidence of post-operative acute rhinosinusitis relative to treatment assignment | Post-op through week 16 post-FESS

SECONDARY OUTCOMES:
Assess week 16 post-FESS Sino-Nasal Outcome Test-22 (SNOT-22) group scores change from baseline relative to treatment assignment | Week 16 post-FESS
Assess antibiotic usage relative to treatment assignment | 1 week post-op through week 16

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No